CLINICAL TRIAL: NCT05495230
Title: tOwards a Patient Centred mulTIMorbidity Approach FOR Chronic Disease MAnagement in Primary Care (OPTIMA FORMA) PHASE 3: Cluster Randomized Controlled Evaluation Study
Brief Title: OPTIMA FORMA Phase 3
Acronym: OPTIMAFORMA3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-15788
Record Dates: First submitted 2022-08-02; First posted 2022-08-10 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2023-11

CONDITIONS: Chronic Condition; Chronic Conditions, Multiple
Keywords: Primary care; General practice; Person-centred integrated care
MeSH Terms: conditions — Chronic Disease; Multiple Chronic Conditions

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Other): Practices in the control group provide care as usual, which consists of the SDM programmes according to the national care standards and General Practice guidelines (NHG) for DM2, COPD and CVD. According to these protocolised programmes, patients with COPD, CVD or DM2 visit their general practice at a standard frequency per year (1 - 4 times) and standard monitoring measurements and topics are discussed.
  The practices that are randomised to the control group will not receive any additional training related to this study.
  Interventions: Other: Usual care
- Person-centred integrated care intervention (Experimental): The core of the person-centered and holistic approach is a cyclical process. The practice nurse in the general practice will act as case manager and can consult the general practitioner or other health providers when necessary. The first step in the intervention is assessing the integral health status of the patient (health across multiple domains, including physiological measurements and symptoms of disease), using a (preferably digital) questionnaire at home and physical measurements. The second step is discussing the results with the patient in a semi-structured way. Personal goals are formulated in the third step. In the fourth step, the healthcare professional and patient will choose through shared-decision making the most appropriate interventions and support to achieve these goals, which are documented in a personal healthcare plan. Next, referrals are made if necessary and the treatment is started. An evaluation is planned and carried out, if necessary multiple times.
  Interventions: Behavioral: Person-centred integrated care intervention

INTERVENTIONS:
Behavioral: Person-centred integrated care intervention — See arm description.
  Arms: Person-centred integrated care intervention
Other: Usual care — See arm description.
  Arms: Usual care

SUMMARY:
Chronic diseases and multimorbidity are increasingly prevalent. However, over the last decades, attempts at improving primary care for chronic diseases have been focussed on the management of individual chronic diseases and single disease management (SDM) programs have been implemented in Dutch primary care. This causes multiple problems for patients with one or more chronic diseases, such as negative interaction between treatment of single diseases, high treatment burden, negative patient experiences, lack of attention for problems in other domains of life that may interact with the chronic disease, and difficulties in shared decision making by the use of strict protocols in SDM programs. A person-centred and holistic approach is widely recognized as the solution to the problems observed in chronic disease care. Therefore, we guided three large Dutch primary care cooperatives, who have been organizing SDM programmes on diabetes mellitus type 2 (DM2), COPD, and cardiovascular diseases (CVD) in primary care for the last decades, with the development of a new generic disease management (GDM) programme including a person-centered and holistic approach (CMO 2019-5756). The three primary care cooperatives have recently conducted a pilot study in which we evaluated the feasibility of the programme (CMO 2021-8106) to further optimise its content and procedures. In the coming years, all three primary care cooperatives will gradually implement the optimised programme in all general practices in their regions. In the current study, our aim is to evaluate the effectiveness of the GDM programme on Quadruple Aim outcomes, i.e. patient experiences, population health, health care provider experiences, and cost effectiveness. We will conduct a cluster randomized controlled trial in the three primary care cooperatives with a follow-up of 12 months. Fifteen practices will be randomised to either care as usual according to the current SDM programmes, or to the GDM programme including a person-centered and holistic care approach. Approximately 40 patients per practice with DM2, COPD and/or CVD will be recruited.

DETAILED DESCRIPTION:
Rationale: Chronic diseases and multimorbidity are increasingly prevalent. However, over the last decades, attempts at improving primary care for chronic diseases have been focussed on the management of individual chronic diseases and single disease management (SDM) programs have been implemented in Dutch primary care. This causes multiple problems for patients with one or more chronic diseases, such as negative interaction between treatment of single diseases, high treatment burden, negative patient experiences, lack of attention for problems in other domains of life that may interact with the chronic disease, and difficulties in shared decision making by the use of strict protocols in SDM programs. A person-centred and holistic approach is widely recognized as the solution to the problems observed in chronic disease care. Therefore, we guided three large Dutch primary care cooperatives, who have been organizing SDM programmes on diabetes mellitus type 2 (DM2), COPD, and cardiovascular diseases (CVD) in primary care for the last decades, with the development of a new generic disease management (GDM) programme including a person-centered and holistic approach (CMO 2019-5756). The three primary care cooperatives have recently conducted a pilot study in which we evaluated the feasibility of the programme (CMO 2021-8106) to further optimise its content and procedures. In the coming years, all three primary care cooperatives will gradually implement the optimised programme in all general practices in their regions.

Objective: In the current study, our aim is to evaluate the effectiveness of the GDM programme on Quadruple Aim outcomes, i.e. patient experiences, population health, health care provider experiences, and cost effectiveness.

Study design: we will conduct a cluster randomized controlled trial in the three primary care cooperatives with a follow-up of 12 months. Fifteen practices will be randomised to either care as usual according to the current SDM programmes, or to the GDM programme including a person-centered and holistic care approach. Approximately 40 patients per practice with DM2, COPD and/or CVD will be recruited.

Study population: all patients with DM2, COPD and/or CVD who currently receive SDM according to the SDM programmes of the participating primary care cooperatives are eligible to participate.

Intervention: a GDM programme including person-centered and holistic care. This programme will replace the SDM programmes for DM2, COPD and CVD that are currently used in the participating primary care cooperatives.

Main study parameters/endpoints: effectiveness will be evaluated by Quadruple Aim outcomes at baseline, at 6 months, and at 12 months follow-up by comparing changes in the intervention group with the comparator group. Patient experiences will be measured with the P3CEQ questionnaire. Population health will be measured with the PROMIS Global-10 questionnaire. Self-management will be measured with the Patient Activation Measure (PAM) score. Healthcare professional experiences will be measured with the MASGZ and the COPILOT questionnaire. Data for calculating costs and conducting a cost-effectiveness analyses will be measured by the Medical Consumption questionnaire and the EQ-5D questionnaire and by process outcomes such as the number and type of consultations and referrals, and duration of consultations from the Electronical Medical Files. At 12 months, a purposive sample of patients and professionals will participate in focus group interviews to collect information on experiences and facilitators and barriers for further implementation. Also, the competences needed by the healthcare professionals to provide personalised and integrated chronic care will be explored.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

* The intervention has been developed by the three primary care cooperatives in close collaboration with their healthcare professionals and their patient panels and with the guidance of our research group. Also, input from the Dutch College of General Practitioners (NHG) and from InEen, the branch organisation for primary care cooperatives, has been obtained to ensure that the intervention will suit their vision and future plans for reorganising Dutch primary care chronic disease management. The intervention is also in line with current movements in healthcare, such as the Positive Health concept.
* All three primary care cooperatives are intending to gradually implement the intervention throughout their regions in the upcoming years. Thus, the GDM programme will be implemented and will replace current SDM, even without the current cluster RCT as proposed in this study protocol.
* The burden and risks associated with the intervention are negligible and comparable with the usual care, i.e. the current SDM programmes.
* Patients in the control group will continue with their care as usual, i.e. single chronic disease management according to the protocols of the SMD programmes that have been used in the participating cooperatives since the last decade.
* The additional burden or risk associated with participation in this study is negligible. After written informed consent, patients in both groups will fill in a digital or paper questionnaire at baseline, 6 months, and 12 months. Estimated time to fill in the questionnaire is 20 minutes. A purposive sample of approximately 15 patients will participate in focus-groups interviews at the end of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in any of the single disease management programmes (usual care) for DM2, COPD, asthma or CVD.

Exclusion Criteria:

* Limited life expectancy (less than 3 months)
* Unable to speak or read the Dutch language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 842 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Composite score HRQoL & patient-experienced quality of healthcare | 12 months
  % difference between intervention group and control group of dichotomous composite score ( yes / no MCID improvement in health-related quality of life or quality of healthcare), which is based on the scores of PROMIS dimensions (GPH, GPM) and the P3CEQ-score.

SECONDARY OUTCOMES:
Global Physical Health | Baseline, 6 months, 12 months
  Physical aspect of health-related quality of life as measured by the PROMIS-Global 10 instrument (T-scores; higher T-score indicates better physical aspect of HrQoL)
Global Mental Health | Baseline, 6 months, 12 months
  Mental aspect of health-related quality of life as measured by the PROMIS-Global 10 instrument (T-scores; higher T-score indicates better mental aspect of HrQoL)
Patient-experienced quality of care | Baseline, 6 months, 12 months
  Person-centredness of care as measured by the Person Centred Coordinated Care Experience Questionnaire (P3CEQ) instrument; minimum score 0, maximum score 30, higher score equals better P3CE.
Patient activation as measured by PAM | Baseline, 6 months, 12 months
  Patient activation as measured by the Patient Activation Measure instrument; minimum 0, maximum 100, higher score equals better patient activation.
Health-related quality of life as measured by the EQ-5D-5L instrument | Baseline, 6 months, 12 months
  Health-related quality of life as measured by the EQ-5D-5L instrument; minimum 0, maximum 1, higher score equals better HrQoL
Health care use according to patient | Baseline, 3 months, 6 months, 9 months, 12 months
  Health care use (number of consultations, number of hospital visits) according to Medical Consumption Questionnaire
BMI | Baseline, 6 months, 12 months
  Combined length and weight according to practice data
HbA1c | Baseline, 6 months, 12 months
  According to practice data
Blood glucose | Baseline, 6 months, 12 months
  According to practice data
Blood LDL-cholesterol | Baseline, 6 months, 12 months
  According to practice data
Systolic and diastolic blood pressure | Baseline, 6 months, 12 months
  According to practice data
Positive affect of healthcare providers | Baseline, 6 months, 12 months
  Satisfaction with job according to selection of MAS-GZ instrument (minimum 8, maximum 40, higher score indicates higher positive affect)
Experience of healthcare providers | Baseline, 6 months, 12 months
  Satisfaction with job according to selection of CO-PILOT instrument (minimum 1, maximum 10, higher score is better experience of healthcare providers)

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-22): https://cdn.clinicaltrials.gov/large-docs/30/NCT05495230/Prot_SAP_000.pdf